CLINICAL TRIAL: NCT06425757
Title: Study on Pharmacokinetics of Single Injection of Ciprofol in Patients With Moderate to Severe Hypoproteinemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xie Kangjie (Other)
Responsible Party: Sponsor-Investigator, Xie Kangjie, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-2024-315(IIT)
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Hypoproteinemia; Pharmacokinetics; Ciprofol
MeSH Terms: conditions — Hypoproteinemia | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Severe Hypoproteinemia (Other): Blood albumin concentration≤30g/L
  Interventions: Drug: ciprofol
- Moderate Hypoproteinemia (Other): Blood albumin concentration 30g/L-40g/L
  Interventions: Drug: ciprofol
- Normal plasma albumin (Other): Blood albumin concentration >40g/L
  Interventions: Drug: ciprofol

INTERVENTIONS:
Drug: ciprofol — Patients who intended to undergo elective surgery under general anesthesia were induced by a single intravenous injection of 0.3mg/kg and ciprofol, and the experimental drug was manually injected by CVC within 30s. 2ml of venous blood was collected before and after administration 0.5min, 1min, 2min, 3min, 5min, 8min, 15min 30min, 1h, 2h and 4h respectively. The concentration of cyclopofol in blood was measured
  Other Names: Si Shuning

SUMMARY:
Blood concentrations of Ciprofol were measured at different time points after single injection in patients with hypoproteinemia

DETAILED DESCRIPTION:
This study was a single-center, interventional clinical study. Patients with different plasma albumin levels were selected before surgery and induced by a single injection of Ciprofol at a depth of 0.3 mg/kg. 2ml of venous blood was collected before and 0.5, 1, 2, 3, 5, 8, 15, 30min, 1h, 2h and 4h after administration. The pharmacokinetics of Ciprofol were studied by measuring the concentration of Ciprofol in blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe hypoproteinemia (albumin < 30g/L, protein detection time uniformly within three days before surgery）
* Weight greater than 45kg, BMI20-24
* The ASA rating is Class I or Class II

Exclusion Criteria:

* Severe liver dysfunction
* Severe renal dysfunction
* Patients with ASA grade III and above
* Known allergy to eggs, soy products, opioids and their relief drugs, propofol
* Emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Blood concentrations at different time points after a single injection | Before administration, after administration 0.5 minute, 1 minute, 2 minutes, 3 minutes, 5 minutes, 8 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours
  Blood concentration of ciprofol

SECONDARY OUTCOMES:
Onset time of ciprofol in patients with hypoproteinemia | Day 1
  The time it takes for the blood concentration of a drug to reach the clinically active concentration level from zero
Effect time of ciprofol in patients with hypoproteinemia | Day 1
  From the time the drug was administered to the time the patient lost consciousness

CONTACTS AND LOCATIONS:
Overall Officials: XIE Kangjie, doctoral, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejang, China